CLINICAL TRIAL: NCT04982939
Title: Efficacy and Safety of Peri-operative Sintilimab in Combination With SOX in Resectable Locally Advanced Gastric Cancer: a Multiple-center Open-label Randomized Phase II Trial.
Brief Title: Peri-operative Sintilimab in Combination With SOX in Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERSIST
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-07

CONDITIONS: Gastric Cancer; Perioperative; Sintilimab
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group-Sintilimab in combination with SOX (Experimental): Preoperative treatment: three cycles of sintilimab in combination with SOX. Radical gastrectomy and lymphadenectomy (D2). Postoperative treatment: five cycles of SOX, Sintilimab up to one year.
  Interventions: Drug: Sintilimab; Drug: S-1; Drug: Oxaliplatin
- Active Comparator-SOX (Active Comparator): Preoperative treatment: three cycles of SOX. Radical gastrectomy and lymphadenectomy (D2). Postoperative treatment: five cycles of SOX.
  Interventions: Drug: S-1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Sintilimab — Sintilimab, 200mg IV d1 Q3W
  Other Names: IBI308
  Arms: Experimental Group-Sintilimab in combination with SOX
Drug: S-1 — S-1, 40-60mg BID d1-14 Q3W
Drug: Oxaliplatin — Oxaliplatin，130mg/m2 d1 Q3W

SUMMARY:
To evaluate efficacy and safety of peri-operative sintilimab in combination with SOX in resectable locally advanced gastric or gastroesophageal junction adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years old ≤ age ≤ 75 years old
* ECOG PS score 0-1
* Treatment naive patients diagnosed as gastric adenocarcinoma or gastroesophageal junction adenocarcinoma by histopathology
* No known HER2-positive status;
* Clinical stage Ⅱ, Ⅲ (T1-4a N+ M0, T3-4a N0 M0, AJCC 8th)
* The research center and the surgeon can complete D2 radical gastrectomy
* Physical condition and organ function allow for larger abdominal surgery
* Sufficient organ and bone marrow function, which is defined as follows:

  1. Blood routine: absolute neutrophil count (ANC)≥1.5×109/L; platelet count (PLT)≥100×109/L; hemoglobin content (HGB)≥9.0 g/dL.
  2. Liver function: Patients without liver metastasis require serum total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ×ULN;
  3. Renal function: Creatinine clearance rate (Ccr) ≥50 mL/min (calculated by Cockcroft/Gault formula):

     1. Female: Ccr= (140-years old) x weight (kg) x 0.85/(72 x serum creatinine (mg/dL))
     2. Male: Ccr= (140-years old) x weight (kg) x 1.00/(72 x serum creatinine (mg/dL))
  4. The coagulation function is adequate, defined as the international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; if the subject is receiving anticoagulation therapy, as long as the PT is within the proposed range of anticoagulation drugs
* LVEF≥50%;
* Agree and be able to comply with the plan during the research period;
* Provide written informed consent before entering the study screening, and the patient has understood that participants can withdraw from the study at any time during the study without any loss;

Exclusion Criteria:

* Complicated with upper gastrointestinal obstruction/bleeding or abnormal digestive function or malabsorption syndrome;
* Complicated with severe uncontrolled concurrent infection or other severe uncontrolled concomitant disease, moderate or severe renal injury;
* Received previous anti-tumor therapy, including chemotherapy, radiotherapy, targeted therapy or immunotherapy, etc.;
* Suffered from other malignant tumors in the past 5 years (except basal cell or squamous cell carcinoma, superficial bladder cancer, cervical cancer in situ or breast cancer);
* Uncontrollable pleural effusion, pericardial effusion or ascites;
* Suffered from severe cardiovascular disease within 12 months before enrollment, such as symptomatic coronary heart disease, congestive heart failure ≥ Grade II, uncontrolled arrhythmia, and myocardial infarction;
* Allergic reactions to the drugs used in this study;
* Use steroids or other systemic immunosuppressive therapies 14 days before enrollment;
* Patients who received study drug treatment within 4 weeks before enrollment (participate in other clinical trials);
* Active autoimmune diseases;
* History of primary immunodeficiency;
* Have used immunosuppressive drugs within 4 weeks before the first dose of study treatment, excluding nasal spray, inhaled or other local glucocorticoids or physiological doses of systemic glucocorticoids (that is, no more than 10 mg/day Pred nisone or other glucocorticoids in equivalent doses), or use hormones to prevent allergy to contrast agents;
* Within 4 weeks before the first dose of study treatment or plan to receive live attenuated vaccine during the study period;
* Known to have active tuberculosis;
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
* HIV antibody positive, active hepatitis B or C (HBV, HCV);
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-06-21 (Estimated); Study Completion 2024-06-21 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | up to 8 weeks after surgery
  Pathological complete response (pCR) rate is defined as the proportion of participants whose tumor in the stomach and lymph node completely disappeared, as determined by a pathologist.

SECONDARY OUTCOMES:
Tumor down-staging rate | up to 8 weeks after surgery
  Tumor down-staging is defined as any stage reduction between clinical and pathologic stage
Major pathological response (MPR) rate | up to 8 weeks after surgery
  Major pathological response (MPR) rate is defined as the proportion of participants whose percentage of residual tumor in the stomach and lymph node decreased to < 10%, as determined by a pathologist.
3 years disease-free survival (DFS) rate | up to 4 years
  3 years disease-free survival (DFS) rate is defined as proportion of participants who have no recurrence or metastasis after 3 years of radical treatment
5 years overall survival (OS) rate | up to 6 years
  5 years overall survival (OS) rate is defined as proportion of participants who survived 5 years after radical treatment
Adverse event | up to 30 days after last treatment administration
  All grades of adverse events, all grades of treatment related adverse events, serious of adverse events
Overall response rate ( ORR) | up to 30 days after last preoperative treatment administration
  Overall response rate ( ORR) is defined as proportion of participants who have a best response of CR or PR
Disease Control Rate (DCR) | up to 30 days after last preoperative treatment administration
  Disease Control Rate (DCR) is defined as proportion of participants who have a best response of CR、PR or SD

CONTACTS AND LOCATIONS:
Overall Officials: Han Liang, PhD., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Xuewei Ding, PhD., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China